CLINICAL TRIAL: NCT02466399
Title: An Open-label Comparison of the Safety and Efficacy of Subconjunctival Liposomal Latanoprost (POLAT-001) to Latanoprost Ophthalmic Solution in Patients With Ocular Hypertension and Primary Open Angle Glaucoma
Brief Title: POLAT-001 Compared to Latanoprost Ophthalmic Solution in Patients With Ocular Hypertension and Open-angle Glaucoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peregrine Ophthalmic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LipoLat-CS202
Record Dates: First submitted 2015-05-27; First posted 2015-06-09 (Estimated); Results first posted 2020-11-16 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-09

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- POLAT-001 (Experimental): Latanoprost liposome ophthalmic injection
  Interventions: Drug: POLAT-001
- Latanoprost ophthalmic solution (Active Comparator): latanoprost ophthalmic solution 0.005%
  Interventions: Drug: Latanoprost ophthalmic solution

INTERVENTIONS:
Drug: POLAT-001 — Subconjunctival injection
  Arms: POLAT-001
Drug: Latanoprost ophthalmic solution — Latanoprost ophthalmic solution q.d., evening
  Arms: Latanoprost ophthalmic solution

SUMMARY:
This is an open-label, randomized, multi-center, active-controlled parallel-comparison of POLAT-001 to latanoprost ophthalmic solution in patients with ocular hypertension and primary open-angle glaucoma.

ELIGIBILITY:
Inclusion Criteria:

1. 18 year of age or greater.
2. Diagnosis of primary open angle glaucoma (OAG) or ocular hypertension (OHT).
3. Unmedicated (post-washout) intraocular pressure (IOP) ≥ 24 mm Hg at 2 eligibility visits (0800 hr), 2-7 days apart. If both eyes meet the IOP criteria, the eye with the higher IOP at Visit 1 will be designated as the study eye. If IOP in both eyes is the same, the right eye will be designated as the study eye. Note that both eyes will be treated.
4. Corrected visual acuity at Visit -1 in each eye +1.0 logarithm of minimum angle of resolution (logMAR) or better by Early Treatment of Diabetic Retinopathy Study (ETDRS) in each eye (equivalent to 20/200).
5. Able and willing to give signed informed consent and follow study instructions.
6. Subjects must have a documented history of ≥ 20% IOP reduction O.U. using any topical ocular prostaglandin/prostamide ocular hypotensive medication.

Exclusion Criteria:

Ophthalmic

1. Glaucoma: pseudoexfoliation or pigment dispersion component, history of angle closure or narrow angles judged to be occludable by the investigator. Note: Previous laser peripheral iridotomy is NOT acceptable.
2. IOP > 36 mm Hg in either eye at any pre-randomization study visit.
3. Known corticosteroid-responder as judged by investigator.
4. Known hypersensitivity to any component of the Investigational Product formulation (benzalkonium chloride, etc.), fluoroquinolone ophthalmic solution, or topical anesthetics, Povidone Iodine antiseptic, or diagnostic eye drops.
5. Previous glaucoma intraocular surgery or glaucoma laser procedures in either eye.
6. Refractive surgery in either eye .
7. Ocular trauma, extraocular or intraocular surgery or laser treatment within the past six months in either eye.
8. Evidence of ocular infection, inflammation, clinically significant blepharitis or conjunctivitis at baseline (Visit 1), or a history of herpes simplex keratitis in either eye. Note: mild blepharitis, allergy and dry eye is acceptable.
9. Ocular medication of any kind within 30 days of Visit 1 in either eye, with the exception of a) ocular hypotensive therapy (which must be washed out according to the provided schedule), b) lid scrubs (which may be used prior to, but not after Visit 1) or c) lubricating drops for dry eye (which may be used throughout the study).
10. Clinically significant ocular disease (e.g. uveitis, severe keratoconjunctivitis sicca) in either eye which might interfere with the study, including glaucomatous damage so severe that washout of ocular hypotensive medications for one month is not judged safe by the investigator (i.e., cup-disc ratio > 0.8).
11. Central corneal thickness greater than 600 µm in either eye.
12. Any ocular abnormality preventing reliable applanation tonometry of either eye.
13. Significant media opacity in either eye that would exclude adequate posterior segment examination
14. Contraindications to pupil dilation in either eye.
15. Unwillingness to accept known adverse events of latanoprost such as eyelid and/or iris pigmentation, eyelash growth, etc.
16. History of macular edema, including cystoid macular edema, or current or recent (6 months) uveitis.
17. Planned intraocular surgery in either eye during study participation

    Systemic:
18. Clinically significant abnormalities (as determined by the treating physician) in laboratory tests at screening.
19. Known hypersensitivity or systemic contraindication to latanoprost or components of study medication.
20. Clinically significant systemic disease (e.g., myasthenia gravis, hepatic, renal, endocrine or cardiovascular disorders), which might interfere with the study.
21. Participation in any investigational study within 30 days prior to baseline.
22. Changes of systemic medication that could have a substantial effect on IOP within 30 days prior to screening, or anticipated during the study.
23. Any individual the investigator believes might suffer physical or mental harm by participating in this trial. Due to the current status of the preclinical safety program, women of childbearing potential who are pregnant, nursing, planning a pregnancy, or not using a medically acceptable form of birth control. An adult woman is considered to be of childbearing potential unless she is one year post-menopausal or three months post-surgical sterilization. All females of childbearing potential must have a negative urine pregnancy test result at the Visit 1 examination and must agree to use an acceptable method of contraception during the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-07; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tina T Wong, MD, Ph.D., Study Director — Peregrine Ophthalmic
Locations (1):
- Professional Research Network, Goose Creek, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | POLAT-001 | Latanoprost Ophthalmic Solution
Started | 53 | 27
Completed | 51 | 27
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Early exit due to family emergency | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | POLAT-001 | Latanoprost Ophthalmic Solution | Total
Number analyzed (Participants) | 53 | 27 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (9.39) | 63.1 (11.69) | 63.9 (10.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 12 | 44
  Male | 21 | 15 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 7 | 21
  Not Hispanic or Latino | 39 | 20 | 59
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 5 | 14
  White | 43 | 22 | 65
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Intraocular Pressure Between Two Measures- Baseline and 3 Months
Description: The mean change from baseline intraocular pressure at 3 months (0800 hrs)
Time Frame: 3 months
Population: Per protocol
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | POLAT-001 | Latanoprost Ophthalmic Solution
Number analyzed (Participants) | 45 | 27
mmHg | -2.3 (4.6) | -6.4 (2.9)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | POLAT-001 | Latanoprost Ophthalmic Solution
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/27
Serious Adverse Events (participants affected / at risk) | 1/53 | 0/27
Other Adverse Events (participants affected / at risk) | 14/53 | 1/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | POLAT-001 (N=53) | Latanoprost Ophthalmic Solution (N=27)
bone and bladder cancer (Renal and urinary disorders) | 1 (1) | 0 (0) — Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Bladder cancer)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | POLAT-001 (N=53) | Latanoprost Ophthalmic Solution (N=27)
Conjunctival haemorrhage (Eye disorders) | 14 (27) | 0 (0)
Foreign body sensation in eyes (Eye disorders) | 9 (9) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 7 (7) | 0 (0)
Instillation site erythema (Eye disorders) | 3 (3) | 0 (0)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If multi-center study publication not published within two (2) years after the completion of the Study at all sites, Investigator may publish the results of the Study obtained by Investigator with 60 days notice to Sponsor